CLINICAL TRIAL: NCT01724177
Title: A Phase 2, Multicenter, Single-arm, Open-label Study to Evaluate the Safety and Efficacy of Lenalidomide in Patients With Relapsed or Recurrent Adult T-cell Leukemia-lymphoma
Brief Title: A Phase 2 Study of Lenalidomide in Patients With Relapsed or Recurrent Adult T-cell Leukemia-lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-ATLL-002
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-03

CONDITIONS: Adult T-Cell Leukemia-Lymphoma
Keywords: Lenalidomide; ATL; ATLL
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide 25mg by mouth (PO) daily until progressive disease or unacceptable toxicity
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 25 mg of Lenalidomide administered orally once daily
  Other Names: Revlimid

SUMMARY:
To evaluate the efficacy of lenalidomide in patients with Adult T-cell Leukemia-lymphoma (ATL) who have previously received chemotherapy for ATL.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign the informed consent
* Aged 20 years or older (at the time of signing the informed consent)
* Have a documented diagnosis of either: acute-, lymphoma-, or unfavorable chronic-type adult T-cell leukemia-lymphoma
* Have received ≥1 prior anti-adult T-cell leukemia-lymphoma therapy, have achieved stable disease or better on their immediately prior therapy and have relapsed or progressed at the time of obtaining signed informed consent
* Subjects for whom at least 1 measurable lesion (measurable lesion of computed tomography scan, peripheral blood or skin lesion) is confirmed in the lesion assessment before registration
* Have an Eastern Cooperative Oncology Group performance status of 0 to 2 at registration
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must agree to comply to Lenalidomide Pregnancy Prevention Risk Management Plan

Exclusion Criteria:

* Have a history of central nervous system involvement or present with central nervous system symptoms, and are diagnosed with central nervous system lymphoma by cerebrospinal fluid cytology examination, head computed tomography scan or brain magnetic resonance imaging during the screening
* Are pregnant or lactating
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study. Examples of such medical condition are, but are not limited to, as follows:

  * Uncontrolled diabetes mellitus as defined by the investigator or sub-investigator
  * Chronic congestive heart failure (New York Heart Association Class III or IV)
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction (within 6 months before starting the study drug)
  * Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia (subjects with controlled atrial fibrillation that is asymptomatic are eligible for this study)
  * Major surgery within 28 days of the start of study treatment
* Exhibit grade 4 neurological disorders
* Patients who are at a high risk for a thromboembolic event and are not willing to take venous thromboembolic prophylaxis.
* Develop active tuberculous disease, herpes simplex, systemic mycosis, or other active infections requiring systemic administration of antibiotics, antiviral agents, or antifungal drugs
* Known human immunodeficiency virus positivity
* Have hepatitis B surface antigen-positive, or hepatitis C virus anti-body positive. In case hepatitis B core antibody and/or hepatitis B surface antibody is positive even if hepatitis B surface antigen-negative, a hepatitis B virus deoxyribonucleic acid test should be performed and if positive the subject will be excluded
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
* Have a history of allogenic stem cell transplantation
* Have received autologous stem cell transplantation within 12 weeks (84 days) of the start of study treatment
* Have previously used lenalidomide
* Have a history of desquamating (blistering) rash while taking thalidomide
* Have received any investigational drugs (unapproved drugs in Japan) within 4 weeks (28 days) of the start of study medication
* Have received any antibody agents within 12 weeks (84 days) of the start of study medication
* Have received chemotherapeutic agents or immunomodulatory drugs for the treatment of adult T-cell leukemia-lymphoma within 4 weeks (28 days) of the start of study treatment
* Have received radiotherapy within 4 weeks (28 days) of the start of study treatment
* Have a history or complication of another malignant tumor other than adult T-cell leukemia-lymphoma and the following malignant tumors, unless the patients have been free of the disease for 5 years or longer

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * Cervical carcinoma in situ
  * Carcinoma in situ of the breast
  * An incidental histological finding of prostate carcinoma (TNM stage T1a or T1b)
  * Early-stage gastric cancer treated with endoscopic mucosal resection or endoscopic submucosal dissection
* Have had any of the following abnormal measurements at screening performed within 1 week (7 days) prior to the registration;

  * Neutrophil count: < 1,200/µL
  * Platelet count: < 75,000/µL
  * Serum aspartate aminotransferase/glutamyl oxaloacetic transaminase or alanine aminotransferase/glutamyl pyruvic transaminase: > 3 times the upper limit of normal
  * Bilirubin level: > 1.5 times the upper limit of normal
  * Creatinine clearance: < 60 mL/min
* Any condition that confounds the ability to interpret data from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2014-11-20 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sasaki, Study Director — Celgene K.K.
Locations (18):
- Japan (18):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tohoku University Hospital, Sendai, Miyagi
  - Sasebo City General Hospital, Sasebo, Nagasaki
  - Heart Life Hospital, Nakagami, Okinawa
  - Shimane University Hospital, Izumo, Shimane
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Imamura Bunin Hospital, Kagoshima
  - Kagoshima University Medical and Dental Hospital, Kagoshima
  - National Hospital Organization Kagoshima Medical Center, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Oita Prefectual Hospital, Ōita
  - National Cancer Center Hospital, Tokyo

REFERENCES:
- [Result] Ishida T, Fujiwara H, Nosaka K, Taira N, Abe Y, Imaizumi Y, Moriuchi Y, Jo T, Ishizawa K, Tobinai K, Tsukasaki K, Ito S, Yoshimitsu M, Otsuka M, Ogura M, Midorikawa S, Ruiz W, Ohtsu T. Multicenter Phase II Study of Lenalidomide in Relapsed or Recurrent Adult T-Cell Leukemia/Lymphoma: ATLL-002. J Clin Oncol. 2016 Dec;34(34):4086-4093. doi: 10.1200/JCO.2016.67.7732. Epub 2016 Sep 30. PMID 27621400

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included Japanese participants with relapsed or recurrent adult T-cell leukemia (ATL) who had previously received anti- ATL chemotherapy and who were categorized as having acute-lymphoma or unfavorable chronic-type ATL.
Groups:
- Lenalidomide: Lenalidomide 25 mg administered by mouth (PO) once daily (QD) until progressive disease or unacceptable toxicity
Period: Overall Study
Arm/Group | Lenalidomide
Started | 26
Safety Population | 26 (Safety Population includes participants who received at least one dose of lenalidomide)
Completed | 0
Not Completed | 26
Not completed — Adverse Event | 8
Not completed — Progressive disease or Relapsed Disease | 16
Not completed — Nervous participant | 1
Not completed — Serious Adverse Event Related | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population consisted of all participants enrolled independent of whether they received study treatment or not.
Groups:
- Lenalidomide: Lenalidomide 25 mg administered orally once daily (QD) until progressive disease or unacceptable toxicity.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (7.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a subject's disease is progressing, assess how the disease affects the daily living activities of the subject and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity) Population: Intent to Treat population was defined as all participants who were enrolled in this study independent of whether they received lenalidomide or not.
  Participants
    0 = Fully Active | 13
    1 = Restrictive but Ambulatory | 9
    2 = Ambulatory but Unable to Work | 4
    3 = Limited Self-Care | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Complete Response, Unconfirmed Complete Response, or Partial Response as Assessed by the Efficacy-Safety Evaluation Committee (ESEC)
Description: ORR is a Complete Response (CR) + Complete Response unconfirmed (CRu) + Partial Response (PR). A CR requires that target lesions have regressed to normal; nodal non-target lesions have regressed to normal; extranodal non-target lesions have disappeared; hepatomegaly/splenomegaly has disappeared; skin findings are GR 0; peripheral blood is normal; Bone marrow (BM) infiltration is negative and no new lesions. A CRu requires the sum of the product diameters (SPD) of target lesions have decreased by at least 75% from baseline; nodal non-target lesions have regressed to normal size; extranodal non-target lesions have disappeared; hepatomegaly/splenomegaly has disappeared; skin findings are Grade 0; peripheral blood is normal; BM infiltration is "negative" and no new lesions. A PR requires the SPD of target lesions has decreased by at least 50% from baseline; all nodal non-target lesions have regressed to normal or show no increase in size; all extranodal non-target lesions have disappeared
Time Frame: From day 1 of study treatment to date of first documented CR, CRU or PR; Up to data cut-off date of 19 May 2017; maximum study duration was 134.1 weeks
Population: The Efficacy Evaluable (EE) population consisted of all participants who met basic protocol requirements (all eligibility criteria) and were evaluated after receiving at least one dose of lenalidomide
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
percentage of participants | 42.3 [23.352 to 63.082]
Statistical Analysis 1: Comparison: Lenalidomide; Test type: Superiority or Other; p < 0.0001, Exact Test — A one sample binomial one sided exact test for the ORR (CR, CRu, or PR) was performed to provide the p-value (significance level: 0.05). The hypotheses of interest: H0: ORR ≤ 5% versus H1: ORR > 5%

2. Secondary Outcome: Kaplan Meier Estimate of Progression Free Survival (PFS) as Assessed by the ESEC
Description: PFS was defined as the time from the first dose of study treatment to progressive disease (PD) or death due to any cause on study or within 28 days after study discontinuation, whichever occurred earlier.
Time Frame: From day 1 of study treatment to the date of disease progression; up to data cut date of date of 19 May 2017; maximum study duration was 134.1 weeks
Population: The EE population consisted of all participants who met basic protocol requirements (all eligibility criteria) and were evaluated after receiving at least one dose of lenalidomide
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
weeks | 16.30 [8.100 to 24.000]

3. Secondary Outcome: Kaplan-Meier Estimate of Time to Progression (TTP)
Description: Time to progression was calculated as the time from the first dosing of study treatment to the first documented PD and assessed by the ESEC
Time Frame: From day 1 of study treatment to the date of disease progression; up to data cut date of 19 May 2017; maximum study duration was 134.1 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
weeks | 16.30 [8.100 to 24.000]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment Emergent Adverse Event (TEAE) was defined as any AE occurring on or after the start of study treatment and within 28 days after the last dose. Severity was assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI CTCAE v4.0): Grade 1= Mild Grade 2= Moderate Grade 3= Severe Grade 4= Life-threatening and Grade 5= Death related to AE. Serious AEs (SAEs) were those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From the date of the first dose of study drug up to 28 days after the last dose of study drug; up to data cutoff date of 19 May 2017; maximum treatment duration was 130.1 weeks
Population: Safety population was defined as all participants who received at least one dose of lenalidomide. All safety analyses were based on the safety population.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
participants
  ≥ 1 TEAE | 26
  ≥ 1 TEAE Related to Lenalidomide | 26
  ≥ 1 NCI CTCAE Grade (GR) 3 or Greater TEAE | 25
  ≥ 1 NCI CTCAE ≥ GR 3 TEAE Related to Lenalidomide | 25
  ≥ 1 Serious TEAE | 11
  ≥ 1 Serious TEAE Related to Lenalidomide | 9
  ≥ 1 TEAE Leading to Discontinuation | 8
  ≥ 1 Related TEAE Leading to Discontinuation | 8
  ≥ 1 TEAE Leading to Dose Reduction/Interruption | 17
  ≥ 1 related TEAE Leading to Decrease/Interruption | 17
  ≥ 1 TEAE Resulting in Death | 0

5. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR) for Responders as Assessed by the ESEC
Description: The response duration in participants with an objective response was measured from the date of the first Complete Response or Complete Response unconfirmed or Partial Response to the first date of Relapsed Disease or Progressive Disease (PD). For participants who did not progress during the study, DOR was censored at the last adequate response assessment not showing evidence of PD.
Time Frame: From day 1 of study treatment to first documented response; up to data cut-off date of 19 May 2017; Maximum study duration was 134.1 Weeks
Population: The EE population who had a documented response and consisted of participants who met basic protocol requirements (all eligibility criteria) and were evaluated after receiving at least one dose of lenalidomide
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
weeks | 24.10 [2.000 to NA] — Only one event data observed exceeding the median value, and maximum value was censored data, so the upper bound of confidence interval (CI) could not be estimated

6. Other Pre Specified Outcome: Time to Response
Description: Time to Response was defined as the time from the first dose of study treatment to the initial documented response (CR or CRu, or PR)
Time Frame: as for outcome 5
Population: Participants with a response of PR or better.
Measure: Median (Full Range); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 11
weeks | 8.10 [7.9 to 16.0]

7. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response, Unconfirmed Complete Response (CRu), Partial Response or Stable Disease (SD) as Assessed by the ESEC
Description: The tumor control rate was measured for those with a response of Complete Remission, + CRu, + PR + Stable Disease (SD) in the EE population based on the best response.
Time Frame: as for outcome 5
Population: The EE population with a response (CR, CRu, PR or SD) and consisted of all participants who met basic protocol requirements (all eligibility criteria) and were evaluated after receiving at least one dose of lenalidomide
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
percentage of participants | 73.1 [52.213 to 88.427]

8. Secondary Outcome: Kaplan-Meier Estimate for Overall Survival
Description: Overall Survival was defined as the time from the start of study treatment to the death due to any cause. For participants who were still alive at the time of the data cutoff, survival data were censored at the latest available date the participant was known to be alive.
Time Frame: From Day 1 of study treatment to disease progression or death; up to final data cut-off date of 19 May 2017; maximum surivival time was 197.9 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 26
weeks | 88.10 [43.000 to 109.100]

ADVERSE EVENTS:
Time Frame: From the first day of lenalidomide treatment through 28 days after the last dose of lenalidomide. up to clinical cut-off date of 19 May 2017; maximum duration of study drug was 130.4 weeks
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 22/26
Serious Adverse Events (participants affected / at risk) | 11/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=26)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Enterocolitis infectious (Infections and infestations) | 1
Meningitis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Acute left ventricular failure (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Blood pressure decreased (Investigations) | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis fungal (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=26)
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Neutropenia (Blood and lymphatic system disorders) | 19
Lymphopenia (Blood and lymphatic system disorders) | 18
Anaemia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 13
Leukocytosis (Blood and lymphatic system disorders) | 5
Basophilia (Blood and lymphatic system disorders) | 3
Eosinophilia (Blood and lymphatic system disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9
Hypoproteinaemia (Metabolism and nutrition disorders) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hyperchloraemia (Metabolism and nutrition disorders) | 3
Hypouricaemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
C-reactive protein increased (Investigations) | 11
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 5
Blood urea increased (Investigations) | 5
Blood creatinine increased (Investigations) | 4
Differential white blood cell count abnormal (Investigations) | 3
Glucose urine present (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 3
Blood urine present (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Malaise (General disorders) | 5
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 4
Oedema peripheral (General disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Bradycardia (Cardiac disorders) | 2
Supraventricular extrasystoles (Cardiac disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Phlebitis (Vascular disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Insomnia (Psychiatric disorders) | 3
Hypogammaglobulinaemia (Immune system disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Eosinophil count increased (Investigations) | 2
Basophil count increased (Investigations) | 2
Blood albumin decreased (Investigations) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements varied; the Investigators shall not disclose any material/information disclosed by the Sponsor (Celgene KK) with the clinical trial or information obtained by conducting the clinical trial to third parties without Sponsor's prior written approval.